CLINICAL TRIAL: NCT03537651
Title: A Phase 3, Open-label, Rollover Study to Evaluate the Safety and Efficacy of Long-term Treatment With Tezacaftor in Combination With Ivacaftor in Subjects With Cystic Fibrosis Aged 6 Years and Older, Homozygous or Heterozygous for the F508del-CFTR Mutation
Brief Title: A Study to Evaluate the Safety and Efficacy of Long-term Treatment With TEZ/IVA in CF Participants With an F508del CFTR Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX17-661-116; 2017-002968-40 (EudraCT Number)
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Results first posted 2021-11-26 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor, ivacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TEZ/IVA (Experimental): Part A: Participants weighing less than (<)40 kilograms (kg) at Day 1 received tezacaftor (TEZ) 50 milligrams (mg) once daily (qd)/ivacaftor (IVA) 75 mg every 12 hours (q12h) and the participants weighing greater than or equals to (>=) 40 kg at Day 1 received TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 96 weeks. Doses were adjusted upward for changes in body weight and/or age.
  Part B: Participants weighing <30 kg at Day 1 received TEZ 50 mg qd/IVA 75 mg q12h and the participants weighing >=30 kg at Day 1 received TEZ 100 mg qd/IVA 150 mg q12h in the treatment period up to 192 weeks. Doses were adjusted upward for changes in body weight and/or age.
  Interventions: Drug: TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: TEZ/IVA — Fixed-dose combination tablet for oral administration.
  Other Names: VX-661/VX-770; tezacaftor/ivacaftor
Drug: IVA — Tablet for oral administration.
  Other Names: VX-770; ivacaftor

SUMMARY:
This study evaluates the long-term safety and tolerability of tezacaftor in combination with ivacaftor (TEZ/IVA) in participants with cystic fibrosis (CF) aged 6 years and older, homozygous or heterozygous for the F508del mutation.

ELIGIBILITY:
Inclusion Criteria:

* Completed the Week 24 Visit in Study 113 Part B or the Week 8 Visit in Study 115
* Eligible CFTR Mutation

Exclusion Criteria:

* Pregnant and nursing females
* History of poor compliance with study drug and/or procedures in a previous study as deemed by the investigator
* Ongoing participation in another study with investigational drug

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (55):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours/ Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Johns Hopkins All Children's Hospital Outpatient Care Center, St. Petersburg, Florida
  - Center for Advanced Pediatrics, Atlanta, Georgia
  - St. Luke's CF Center of Idaho, Boise, Idaho
  - Riley Hospital for Children Indiana University Health, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital & Clinics of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Dartmouth Hitchcock Medical Center, Manchester, New Hampshire
  - UBMD Pediatrics/ CF Center of Western New York, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Sanford Children's Speciality Clinic, Sioux Falls, South Dakota
  - Austin Children's Chest Associates, Austin, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Perth Children's Hospital, Nedlands
  - John Hunter Hospital & Hunter Medical Research Institute and John Hunter Children's Hospital, New Lambton
  - Lady Cilento Children's Hospital, South Brisbane
  - The Children's Hospital at Westmead, Westmead
- Belgium (2):
  - Universitair Ziekenhuis Brussel - Campus Jette, Brussels
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Canada (3):
  - British Columbia's Children's Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Centre, Glen Site, Montreal Children's Hospital, Montreal, Quebec
- Juliane Marie Center, Rigshopitalet, Copenhagen, Denmark
- France (2):
  - Groupe Hospitaler Pellegrin, CHU De Bordeaux, Bordeaux
  - Hopital Necker, Enfants Malades, Paris
- Germany (7):
  - Universitaetsklinkum Koeln, CF-Studienzentrum, Cologne
  - Universitätsklinikum Essen, Essen
  - Clinic of J.W. Goethe University, Frankfurt
  - Justus-Leibig-Universitat Zentrum fur Kinderheilkunde und Jugendmedizin, Giessen
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Jena, Mukoviszidose-Zentrum, Jena
  - Universitaetsklinikum Tuebingen Klinik fuer Kinder- und Jugendmedizin, Tübingen
- Ireland (2):
  - Our Lady's Children's Hospital, Dublin
  - University Hospital Limerick, Limerick
- Klinika Mukowiscydozy IMD Oddozial Chorob Pluc Szpzoz IM. Dzieci WarszaWY, Łomianki, Poland
- Switzerland (2):
  - Inselspital - Universitaetsspital Bern, Bern
  - Kinderspital Zuerich, Zurich
- United Kingdom (3):
  - Leeds General Infirmary, Leeds
  - Royal Brompton & Harefield NHS Foundation Trust, Royal Brompton Hospital, London
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Sawicki GS, Chilvers M, McNamara J, Naehrlich L, Saunders C, Sermet-Gaudelus I, Wainwright CE, Ahluwalia N, Campbell D, Harris RS, Paz-Diaz H, Shih JL, Davies JC. A Phase 3, open-label, 96-week trial to study the safety, tolerability, and efficacy of tezacaftor/ivacaftor in children >/= 6 years of age homozygous for F508del or heterozygous for F508del and a residual function CFTR variant. J Cyst Fibros. 2022 Jul;21(4):675-683. doi: 10.1016/j.jcf.2022.02.003. Epub 2022 Feb 18. PMID 35190292
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 parts, Part A and Part B. Participants from Part A also participated in Part B. The Participant flow was planned to be presented for the overall treatment arm.
Pre-assignment Details: This study was conducted in cystic fibrosis (CF) participants aged 6 years or older who participated in parent studies VX15-661-113 Part B (Study 113B; NCT02953314) or VX16-661-115 (Study 115; NCT03559062). Eligible participants from parent studies were enrolled in Study 116.
Groups:
- TEZ/IVA: Part A: Participants weighing less than (<)40 kilograms (kg) at Day 1 received tezacaftor (TEZ) 50 milligrams (mg) once daily (qd)/ivacaftor (IVA) 75 mg every 12 hours (q12h) and the participants weighing greater than or equals to (>=) 40 kg at Day 1 received TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 96 weeks. Doses were adjusted upward for changes in body weight and/or age.
  Part B: Participants weighing <30 kg at Day 1 received TEZ 50 mg qd/IVA 75 mg q12h and the participants weighing >=30 kg at Day 1 received TEZ 100 mg qd/IVA 150 mg q12h in the treatment period upto192 weeks. Doses were adjusted upward for changes in body weight and/or age.
Period: Part A (Up to 96 Weeks)
Arm/Group | TEZ/IVA
Started | 130
113B/116 FAS (All enrolled participants from parent Study 113B who received at least 1 dose of TEZ/IVA in Study 116 and had an eligible genotype.) | 64
113B/116 LCI FAS (All enrolled participants who participated in the LCI sub study in parent Study 113B and received at least 1 dose of TEZ/IVA in Study 116 and had an eligible genotype.) | 30
115/116 FAS (All enrolled participants who were randomized to either TEZ/IVA, IVA or placebo treatment group in parent Study 115 and received at least 1 dose of TEZ/IVA in Study 116 and had an eligible genotype.) | 66
115/116 FAS (TEZ/IVA Group) (All enrolled participants who were randomized to the TEZ/IVA treatment group in parent Study 115 and received at least 1 dose of TEZ/IVA in Study 116 and had an eligible genotype.) | 53
Completed | 69
Not Completed | 61
Not completed — Adverse Event | 2
Not completed — Withdrawal of Consent (not due to AE) | 2
Not completed — Commercial Drug is Available for Participant | 56
Not completed — Other | 1
Period: Part B (Up to 192 Weeks)
Arm/Group | TEZ/IVA
Started | 62 (Out of the 130 participants from Part A, only 62 participants participated in Part B of the study.)
113B/116 FAS (All enrolled participants from parent Study 113B who received at least 1 dose of TEZ/IVA in Study 116 and had an eligible genotype.) | 9
115/116 FAS (All enrolled participants who were randomized to either TEZ/IVA, IVA or placebo treatment group in parent Study 115 and received at least 1 dose of TEZ/IVA in Study 116 and had an eligible genotype.) | 53
Completed | 3
Not Completed | 59
Not completed — Adverse Event | 1
Not completed — Withdrawal of Consent (not due to AE) | 1
Not completed — Commercial Drug is available for Participant | 56
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Baseline is defined as the most recent non-missing measurement (scheduled or unscheduled) collected before the first dose of TEZ/IVA in either the parent study or Study 116. Baseline data is presented for participants who received at least 1 dose of study drug in this study.
Groups:
- TEZ/IVA: Part A: Participants weighing <40 kg at Day 1 received TEZ 50 mg qd/ IVA 75 mg q12h and the participants weighing >= 40 kg at Day 1 received TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 96 weeks. Doses were adjusted upward for changes in body weight and/or age.
  Part B: Participants weighing <30 kg at Day 1 received TEZ 50 mg qd/IVA 75 mg q12h and the participants weighing >=30 kg at Day 1 received TEZ 100 mg qd/IVA 150 mg q12h in the treatment period up to 192 weeks. Doses were adjusted upward for changes in body weight and/or age.
Arm/Group | TEZ/IVA
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The Baseline data were planned to be presented separately for Part A and Part B. Here "Number Analyzed" signifies participants who were evaluable for the specified part of the study.
  years
    Part A | 8.3 (1.7)
    Part B: number analyzed (Participants) | 62
    Part B | 8.3 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented separately for Part A and Part B. Here "Number Analyzed" signifies participants who were evaluable for the specified part of the study.
  Participants
    Part A: Female | 67
    Part A: Male | 63
    Part B: number analyzed (Participants) | 62
    Part B: Female | 35
    Part B: Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented separately for Part A and Part B. Here "Number Analyzed" signifies participants who were evaluable for the specified part of the study.
  Participants
    Part A: Hispanic or Latino | 4
    Part A: Not Hispanic or Latino | 119
    Part A: Not collected per local regulations | 7
    Part B: number analyzed (Participants) | 62
    Part B: Hispanic or Latino | 3
    Part B: Not Hispanic or Latino | 52
    Part B: Not collected per local regulations | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented separately for Part A and Part B. Here "Number Analyzed" signifies participants who were evaluable for the specified part of the study.
  Participants
    Part A: White | 125
    Part A: Black or African American | 1
    Part A: Asian | 1
    Part A: Not collected per local regulations | 2
    Part A: Other | 1
    Part B: number analyzed (Participants) | 62
    Part B: White | 59
    Part B: Black or African American | 1
    Part B: Asian | 0
    Part B: Not collected per local regulations | 2
    Part B: Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 100
Population: Safety Set included all participants who were enrolled and received at least 1 dose of TEZ/IVA in Part A of Study 116.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: TEZ/IVA: Participants weighing <40 kg at Day 1 received TEZ 50 mg qd/IVA 75 mg q12h and the participants weighing >= 40 kg at Day 1 received TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 96 weeks. Doses were adjusted upward for changes in body weight and/or age.
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 130
Participants
  Participants With TEAEs | 129
  Participants With SAEs | 31

2. Secondary Outcome: Part A: Absolute Change in Lung Clearance Index2.5 (LCI2.5) for 115/116 FAS (TEZ/IVA Group)
Description: The LCI2.5 index is the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/40th of its starting values and is calculated by dividing the sum of exhaled tidal breaths (cumulative exhaled volume (CEV)) by simultaneously measured functional residual capacity (FRC). An LCI of 7.5 and below is normal; values greater than 7.5 are abnormal. LCI is able to detect abnormalities in lung function earlier than more traditional modalities such as spirometry.
Time Frame: From Parent Study 115 Baseline at Week 96 (Study 116)
Population: 115/116 Full analysis set (FAS) (TEZ/IVA group) included all enrolled participants who were randomized to the TEZ/IVA treatment group in parent Study 115 and received at least 1 dose of TEZ/IVA in Study 116 and had an eligible genotype. As pre-specified in the SAP, model-based efficacy analysis for participants from parent Study 115 was planned only for the TEZ/IVA treatment group.
Measure: Least Squares Mean (95% Confidence Interval); unit: Index
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 53
Index | -0.95 [-1.38 to -0.52]

3. Secondary Outcome: Part A: Absolute Change in LCI2.5 for 113B/116 LCI FAS
Description: as for outcome 2
Time Frame: From Parent Study 113B Baseline at Week 96 (Study 116)
Population: 113B/116 LCI FAS included all enrolled participants who participated in the LCI sub study in parent Study 113B and received at least 1 dose of TEZ/IVA in Study 116 and had an eligible genotype. As pre-specified in the SAP, only descriptive summary statistics were planned to be reported for the 113B/116 LCI FAS.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 30
Index | -2.04 (1.73)

4. Secondary Outcome: Part A: Absolute Change in Sweat Chloride (SwCl) for 115/116 FAS (TEZ/IVA Group)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Parent Study 115 Baseline at Week 96 (Study 116)
Population: 115/116 FAS (TEZ/IVA group). As pre-specified in the SAP, model-based efficacy analysis for participants from parent Study 115 was planned only for the TEZ/IVA treatment group.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Groups:
- TEZ/IVA: Participants weighing <40 kg at Day 1 received TEZ 50 mg qd/IVA 75 mg q12h and the participants weighing >= 40 kg at Day 1 received TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 96 weeks. Doses were adjusted upward for changes in body weight and/or age.
Arm/Group | TEZ/IVA
Number analyzed (Participants) | 53
millimole per liter (mmol/L) | -13.8 [-17.7 to -9.9]

5. Secondary Outcome: Part A: Absolute Change in SwCl for 113B/116 FAS
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Parent Study 113B Baseline at Week 96 (Study 116)
Population: 113B/116 FAS included all enrolled participants from parent Study 113B who received at least 1 dose of TEZ/IVA in Study 116 and had an eligible genotype.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 64
mmol/L | -16.2 [-21.9 to -10.5]

6. Secondary Outcome: Part A: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score for 115/116 FAS (TEZ/IVA Group)
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with CF. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: From Parent Study 115 Baseline at Week 96 (Study 116)
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 53
units on a scale | 6.4 [3.5 to 9.3]

7. Secondary Outcome: Part A: Absolute Change in CFQ-R Respiratory Domain Score for 113B/116 FAS
Description: as for outcome 6
Time Frame: From Parent Study 113B Baseline at Week 96 (Study 116)
Population: 113B/116 FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 64
units on a scale | 6.0 [1.1 to 10.8]

8. Secondary Outcome: Part A: Absolute Change in Body Mass Index (BMI) for 115/116 FAS (TEZ/IVA Group)
Description: BMI was defined as weight in kilograms (kg) divided by squared height in meters (m^2).
Time Frame: From Parent Study 115 Baseline at Week 96 (Study 116)
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: kilogram per meter square (kg/m^2)
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 53
kilogram per meter square (kg/m^2) | 1.25 [1.00 to 1.49]

9. Secondary Outcome: Part A: Absolute Change in BMI for 113B/116 FAS
Description: BMI was defined as weight in kg divided by m^2.
Time Frame: From Parent Study 113B Baseline at Week 96 (Study 116)
Population: 113B/116 FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 64
kg/m^2 | 1.19 [0.74 to 1.64]

10. Secondary Outcome: Part B: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 192
Population: Safety Set included all participants who were enrolled and received at least 1 dose of TEZ/IVA in Part B of Study 116.
Measure: Count of Participants; unit: Participants
Groups:
- TEZ/IVA: Part B: Participants weighing <30 kg at Day 1 received TEZ 50 mg qd/IVA 75 mg q12h and the subjects weighing >=30 kg at Day 1 received TEZ 100 mg qd/IVA 150 mg q12h in the treatment period up to 192 weeks. Doses were adjusted upward for changes in body weight and/or age
Arm/Group | TEZ/IVA
Number analyzed (Participants) | 62
Participants
  Participants with TEAEs | 53
  Participants with SAEs | 8

ADVERSE EVENTS:
Time Frame: Day 1 Through Safety Follow-up Visit (up to Week 100 for Part A, and up to Week 192 for Part B)
Description: Safety Set included all participants who were enrolled and received at least 1 dose of TEZ/IVA in Study 116.MedDRA version 23.1 applied for Part A, MedDRA version 26.1 applied for Part B.
Groups:
- Part B: TEZ/IVA: Participants weighing <30 kg at Day 1 received TEZ 50 mg qd/IVA 75 mg q12h and the participants weighing >=30 kg at Day 1 received TEZ 100 mg qd/IVA 150 mg q12h in the treatment period up to 192 weeks. Doses were adjusted upward for changes in body weight and/or age.
Arm/Group | Part A: TEZ/IVA | Part B: TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 0/130 | 0/62
Serious Adverse Events (participants affected / at risk) | 31/130 | 8/62
Other Adverse Events (participants affected / at risk) | 128/130 | 49/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: TEZ/IVA (N=130) | Part B: TEZ/IVA (N=62)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cystic fibrosis related diabetes (Congenital, familial and genetic disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Bacterial disease carrier (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 15 | 1
Influenza (Infections and infestations) | 1 | 0
Pertussis (Infections and infestations) | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Bacterial test positive (Investigations) | 3 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Pseudomonas test positive (Investigations) | 0 | 1
Pulmonary function test decreased (Investigations) | 1 | 0
Stenotrophomonas test positive (Investigations) | 1 | 0
Weight gain poor (Metabolism and nutrition disorders) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Personality change (Psychiatric disorders) | 1 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: TEZ/IVA (N=130) | Part B: TEZ/IVA (N=62)
Ear pain (Ear and labyrinth disorders) | 8 | 0
Abdominal pain (Gastrointestinal disorders) | 20 | 6
Abdominal pain upper (Gastrointestinal disorders) | 8 | 1
Constipation (Gastrointestinal disorders) | 10 | 4
Diarrhoea (Gastrointestinal disorders) | 8 | 0
Nausea (Gastrointestinal disorders) | 8 | 3
Vomiting (Gastrointestinal disorders) | 21 | 5
Fatigue (General disorders) | 7 | 0
Pyrexia (General disorders) | 26 | 3
Bacterial disease carrier (Infections and infestations) | 7 | 6
COVID-19 (Infections and infestations) | 0 | 15
Ear infection (Infections and infestations) | 8 | 2
Gastroenteritis (Infections and infestations) | 9 | 2
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 57 | 10
Influenza (Infections and infestations) | 13 | 0
Nasopharyngitis (Infections and infestations) | 24 | 10
Otitis media (Infections and infestations) | 8 | 4
Pharyngitis (Infections and infestations) | 8 | 0
Pharyngitis streptococcal (Infections and infestations) | 8 | 0
Rhinitis (Infections and infestations) | 11 | 4
Tonsillitis (Infections and infestations) | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 31 | 10
Viral upper respiratory tract infection (Infections and infestations) | 10 | 3
Alanine aminotransferase increased (Investigations) | 12 | 2
Aspartate aminotransferase increased (Investigations) | 8 | 2
Bacterial test positive (Investigations) | 19 | 8
Forced expiratory volume decreased (Investigations) | 7 | 7
Pseudomonas test positive (Investigations) | 11 | 2
Staphylococcus test positive (Investigations) | 3 | 4
Headache (Nervous system disorders) | 20 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 73 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 24 | 2
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 24 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 22 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 14 | 3
Rash (Skin and subcutaneous tissue disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT03537651/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT03537651/SAP_001.pdf